CLINICAL TRIAL: NCT01235234
Title: A Phase 3, Randomized, Double-Masked, Placebo-Controlled, Dose-Finding, Parallel-Group Study of the Safety and Efficacy of Daily CF101 Administered Orally in Patients With Moderate-to-Severe Dry Eye Disease
Brief Title: Trial of CF101 to Treat Patients With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-301KCS
Record Dates: First submitted 2010-11-03; First posted 2010-11-05 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry eye disease; KCS; Aqueous Deficient Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CF101 0.1 mg (Experimental): Subjects were randomized to receive CF 101 0.1mg, orally, twice daily for 24 weeks
  Interventions: Drug: CF101
- CF101 1 mg (Experimental): Subjects were randomized to receive CF 101 1.0mg, orally, twice daily for 24 weeks
  Interventions: Drug: CF101
- Placebo (Placebo Comparator): Subjects were randomized to receive matching placebo, orally, twice daily for 24 weeks
  Interventions: Drug: CF101

INTERVENTIONS:
Drug: CF101 — orally q12h
  Other Names: IB-MECA

SUMMARY:
Eligible patients with dry eye will be treated with CF101 or placebo twice daily for 24 weeks. Disease activity will be assessed using evaluations of ocular surface integrity, tear production, and patient symptoms.

DETAILED DESCRIPTION:
Patients will be randomized to receive either CF101 0.1 mg, CF101 1.0 mg, or matching placebo, given orally twice daily (BID) for 24 weeks. A Screening Period of up to 4 weeks that includes a 2-week run-in period will precede a 24-week treatment period, followed by a 2-week follow-up period.

At a Screening Visit, patients will undergo complete medical and ophthalmologic history, medication history, physical examination (including height, weight, sitting blood pressure, pulse rate and temperature), ophthalmic examination, and clinical laboratory tests. Disease activity will be assessed using fluorescein staining, Schirmer test with and without anesthesia, Ocular Surface Disease Index©, and tear break-up time.

Eligible patients will begin a 2-week run-in period during the 4-week screening period, during which time they will be instructed to discontinue use of all topical ophthalmic medications except for REFRESH TEARS® Lubricant Eye Drops. At the Baseline Visit, patients who successfully complete the 2-week run-in period and re-qualify for entry will be randomized to their assigned medication (CF101 0.1 mg, CF101 1.0 mg, or matching placebo) to be taken orally twice daily BID for 24 weeks. Patients will return for assessments and a new supply of study medication at Weeks 2, 4, 8, 12, 16, and 20; at Week 24 for a final on-treatment assessment; and at Week 26 for the 2-week off-treatment follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and over;
* Have a diagnosis of moderate-to-severe Aqueous-Deficient Dry Eye (including Sjögren's Syndrome dry eye), as defined by:

  1. Positive corneal fluorescein staining (FS), defined as a corneal punctate fluorescein staining score of ≥4 in either eye by the National Eye Institute evaluation scale summed over 5 areas each with a 0-3 scoring scale; AND
  2. FS score of ≥2 in at least one corneal region; AND
  3. Schirmer Test (ST) score (without anesthesia) ≥1 mm and < 7 mm/5 min in either eye; AND
  4. OSDI score of ≥20;
* Central corneal FS score of ≥2 in at least 1 eye;
* Willing to use no topical ocular treatments, other than REFRESH® unpreserved artificial tears up to a maximum of 4 times daily, for the duration of the trial (including the 2-week run-in period, the 24-week treatment period and the 2-week follow-up period);
* Willing to forego periocular cosmetic application for the duration of the trial;
* Females of child-bearing potential must have a negative urine pregnancy test at screening and throughout the study, to be eligible for, and continue participation in, the study;
* Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the Investigator (for example oral contraceptive pills plus a barrier method) to be eligible for, and continue participation in, the study;
* Ability to complete the study in compliance with the protocol; and
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Sjögren's Syndrome with significant systemic non-exocrine gland involvement which, in the investigator"s opinion, would interfere with the conduct of the trial;
* Stevens-Johnson Syndrome;
* Use of methotrexate or systemic cyclosporine within the 3 months prior to the Screening Visit;
* of any other disease-modifying anti-rheumatic therapy within 2 months prior to the Screening Visit;
* Use of any anti-rheumatic biological agent within 2 months, or 5 half-lives, whichever is longer, prior to the Screening Visit;
* Use of oral corticosteroids >10 mg prednisone, or equivalent, per day;
* Use of topical steroids within 4 weeks prior to the Screening Visit and for the duration of the study;
* Receipt of topical cyclosporine eye drops within 3 months prior to the Screening Visit and for the duration of the trial;
* Use of oral statin or preparation containing omega-3 fatty acid unless dose has been stable for at least 3 months and will remain so during the course of the trial;
* Presence of chronic ocular disease other than Aqueous-Deficient Dry Eye requiring topical treatment;
* Presence of post-burn ocular injury;
* Ocular herpes simplex virus infection;
* Concomitant use of contact lenses or use within 3 months prior to the Screening Visit;
* Persistent intraocular inflammation or infection;
* Active anterior blepharitis of greater than mild degree, defined as minimal crust at the base of the eyelashes and no signs of inflammation;
* Meibomian gland dysfunction (MGD) of greater than mild degree, defined as mild plugging of the Meibomian glands without lid margin inflammation;
* Surgical occlusion of the lacrimal puncta, including the insertion of punctual plugs, within 3 months of the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2011-07; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma
Locations (1):
- Bnei Zion Medical Center, Haifa, Israel

REFERENCES:
- [Background] Avni I, Garzozi HJ, Barequet IS, Segev F, Varssano D, Sartani G, Chetrit N, Bakshi E, Zadok D, Tomkins O, Litvin G, Jacobson KA, Fishman S, Harpaz Z, Farbstein M, Yehuda SB, Silverman MH, Kerns WD, Bristol DR, Cohn I, Fishman P. Treatment of dry eye syndrome with orally administered CF101: data from a phase 2 clinical trial. Ophthalmology. 2010 Jul;117(7):1287-93. doi: 10.1016/j.ophtha.2009.11.029. Epub 2010 Mar 20. PMID 20304499
- See also: Sponsor — http://www.canfite.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo
Started | 77 | 78 | 81
Completed | 75 | 76 | 80
Not Completed | 2 | 2 | 1
Not completed — Adverse Event | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo | Total
Number analyzed (Participants) | 77 | 78 | 81 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 57 | 56 | 59 | 172
  >=65 years | 20 | 22 | 22 | 64
Age, Continuous [Mean (Full Range); unit: years] | 56.8 [22 to 82] | 54.5 [19 to 90] | 55.1 [20 to 86] | 55.5 [19 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 62 | 71 | 188
  Male | 22 | 16 | 10 | 48
Region of Enrollment [Number; unit: participants]
  Israel | 77 | 78 | 81 | 236

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Complete Clearing of Corneal Staining (i.e., Total Corneal FS Score = 0) at Week 24
Description: Complete clearing of corneal staining by fluorescein staining (FS). The primary efficacy analysis was performed for 1eye (target eye), defined as the eye with the larger corneal FS value at Baseline. If both eyes had the same corneal FS value at baseline, the target eye was considered the eye with the larger central corneal staining value at Baseline. Corneal FS defined as a corneal punctate fluorescein staining score of ≥4 in either eye by the National Eye Institute evaluation scale summed over 5 areas each with a 0-3 scoring scale
Time Frame: 24 weeks
Population: The Number of Subjects Who Achieved Complete Clearing of Corneal Staining in Target Eye Using NRI at 24 weeks (ITT Population)
Measure: Number; unit: participants
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo
Number analyzed (Participants) | 76 | 77 | 76
participants
  Complete clearing of corneal staining in target eye using NRI - YES | 15 | 13 | 21
  Complete clearing of corneal staining in target eye using NRI - NO | 61 | 64 | 55

2. Primary Outcome: Number of Subjects With Adverse Events
Description: Determine the safety of oral CF 101 in this subject population. Adverse Events (AEs) and changes in vital signs, physical examination, clinical laboratory tests (liver, kidney, hematology, chemistry and urinalysis), electrocardiogram (ECG) findings, slit lamp and ophthalmic examination, visual acuity, and intraocular pressure measurements.
Time Frame: 24 weeks
Population: Safety Population - Adverse Events
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo
Number analyzed (Participants) | 77 | 78 | 81
Participants
  Any AEs | 29 | 37 | 29
  Blood and lymphatic system disorders | 1 | 0 | 3
  Cardiac disorders | 4 | 6 | 6
  Ear and labyrinth disorders | 1 | 1 | 0
  Endocrine disorders | 1 | 1 | 0
  Eye disorders | 6 | 8 | 3
  Gastrointestinal disorders | 3 | 5 | 4
  General disorders and administration site conditions | 1 | 4 | 2
  Immune system disorders | 1 | 0 | 2
  Infections and infestations | 3 | 2 | 0
  Investigations | 4 | 9 | 1
  Musculoskeletal and connective tissue disorders | 2 | 5 | 1
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) | 1 | 0 | 1
  Nervous system disorders | 4 | 6 | 4
  Psychiatric disorders | 1 | 1 | 0
  Renal and urinary disorders | 10 | 16 | 11
  Reproductive system and breast disorders | 2 | 3 | 1
  Respiratory, thoracic and mediastinal disorders | 2 | 1 | 7
  Skin and subcutaneous tissue disorders | 2 | 5 | 1
  Vascular disorders | 2 | 4 | 4

3. Secondary Outcome: Number of Subjects Who Achieve an Increase in Schirmer Test Tearing by >9mm Over Baseline
Description: ST wetting increase over Baseline of ≥10 mm with or without anesthesia in either eye at Week 24, using a strip of filter paper placed inside the lower eyelid
Time Frame: 24 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo
Number analyzed (Participants) | 76 | 77 | 76
Participants
  Number of subjects with ST wetting increase over baseline of >=10mm at 24 weeks | 15 | 13 | 13
  Number of subjects without ST wetting increase over baseline of >=10mm at 24 weeks | 61 | 64 | 63

4. Secondary Outcome: Ocular Surface Disease Index
Description: The Ocular Surface Disease Index is assessed on a scale of 0 to 100, with higher scores representing greater disability.
  The subtotal score is based on 12 questions with answers ranging from 0 - "none the time," to 4 - "all of the time."
  The number of questions answered is totaled (0 - 12).
  The OSDI is calculated using the sum of subtotal scores (0-48) multiplied by 25, divided by number of questions answered (0-12). (i.e., if a participant answers all 12 questions with a severe outcome of 4, their respected OSDI = [(4 x 12) x 25] / 12 = [48 x 25] / 12 = 100)
  The outcome measured is the Mean Change from Baseline in Ocular Surface Disease Index at Week 24
Time Frame: 24 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Score on a Scale - OSDI
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo
Number analyzed (Participants) | 76 | 77 | 76
Score on a Scale - OSDI | -24.27 (17.99) | -25.63 (16.77) | -28.70 (19.08)

ADVERSE EVENTS:
Arm/Group | CF101 0.1 mg | CF101 1 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/77 | 0/78 | 1/81
Other Adverse Events (participants affected / at risk) | 9/77 | 13/78 | 9/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 0.1 mg (N=77) | CF101 1 mg (N=78) | Placebo (N=81)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — Bilateral pneumonia
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 — Inflammation of right facial nerve
Cerebral aneurysm ruptured syphilitic (Nervous system disorders) | 1 | 0 | 0 — Left middle cerebral artery bifurcation aneurysm
Endometrial cancer (Reproductive system and breast disorders) | 1 | 0 | 0 — Moderately differentiated endometrioid adenocarcinoma
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 1 — CVA
Type 2 diabetes mellitus (Endocrine disorders) | 1 | 0 | 0 — Diabetes mellitus type II
Hypertension (Vascular disorders) | 1 | 0 | 0 — Iatrogenic orthostatic hypotension remitted
Angina unstable (Cardiac disorders) | 1 | 0 | 0 — Unstable angina
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 0.1 mg (N=77) | CF101 1 mg (N=78) | Placebo (N=81)
Urinary tract infection (Renal and urinary disorders) | 9 | 13 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No